CLINICAL TRIAL: NCT02437864
Title: Effect of Peri-intubation Apneic Oxygenation Via Nasal Cannula on Pediatric Patients' Oxygen Saturation During Airway Management
Brief Title: Apneic Oxygenation During Airway Management in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Codruta Soneru, Assistant Professor, University of New Mexico
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 14-307
Record Dates: First submitted 2015-04-30; First posted 2015-05-08 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baseline Group (No Intervention): Airway management (intubation) undertaken immediately after anesthetic induction, without simultaneous supplemental oxygen via nasal cannula.
- With-Cannula Group (Experimental): Airway management (intubation) undertaken immediately after anesthetic induction, with simultaneous supplemental oxygen via nasal cannula.
  Interventions: Device: Supplemental oxygen via nasal cannula

INTERVENTIONS:
Device: Supplemental oxygen via nasal cannula
  Arms: With-Cannula Group

SUMMARY:
Airway placement after anesthetic induction in pediatric patients is routinely performed at our institution without apneic oxygenation. When intubation is attempted by an inexperienced (learner) provider, the attending physician intervenes if necessary before the patient experiences excessive loss of oxygenation. The investigators plan to institute routine supplemental oxygenation via nasal cannula during this placement. This study will examine the effect of adding apneic oxygenation via nasal cannula on oxygen saturation.

DETAILED DESCRIPTION:
This observational (i.e. nonrandomized) study aims to investigate the effect of a planned practice change; instituting oxygenation via nasal cannula during induction of anesthesia. The use of a nasal cannula during the peri-intubation period is of minimal risk and is not considered a standard of care in pediatric anesthesia. Some providers use it in certain clinical situations, but it is not broadly used and has virtually no pediatric literature to support or refute its use. At our institution, intubation of pediatric patients by inexperienced (learner) providers under expert supervision is routine. The attending physician intervenes if necessary before the patient experiences excessive loss of oxygenation.

Participants will be enrolled in the study once they have entered the pre-operative area and are determined by the attending anesthesiologist to be an eligible study participant. Participants enrolled in the first three months of the study (up to N=200) will be assigned to the baseline condition as described below. Participants enrolled in the second phase of the study (up to N=300) will be assigned to the with-cannula condition described below.

Apneic oxygenation is based on the physiology of the lungs: they absorb a greater volume of oxygen, 250 ml/min in an adult, than the volume of carbon dioxide, 8-20 mL/min, that is released by the lungs, because the majority of carbon dioxide is buffered in the blood stream during apnea. With the imbalanced volumes of absorption and release of gases in the lungs there is a lower than atmospheric pressure in the lungs, creating a passive movement of gases from pharynx to alveoli. If the gas in the pharynx has a significantly higher percentage of oxygen instead of room air at 21% oxygen, a higher amount of oxygen can be passively delivered to the lungs for absorption prolonging the time to hemoglobin desaturation.

For the Baseline Group of this observational (nonrandomized) study, all intubation procedures will be performed as per usual practice. Patients will receive premedication as determined by anesthesiologist/resident/midlevel. Once patients are brought to the operating room and vital signs are being monitored, patients will be preoxygenated via mask per standard of care, with an expired oxygenation concentration minimum of 0.75. Vitals will be recorded at the moment prior to removal of the face mask at the end of the preoxygenation period. Anesthetic induction will be performed with agents and dosages as per the provider's clinical judgment. Airway management consisting of oral endotracheal intubation or laryngeal mask airway insertion will take place. As per standard of care, an attending physician who is expert in pediatric airway management will supervise the procedure and intervene before the patient experiences excessive oxygen desaturation.

For the With-Cannula Group, all of the above steps will be maintained. The sole difference will be nasal cannula placement after induction. It will be set to deliver oxygen at 5 liters per minute. Airway management consisting of oral endotracheal intubation or laryngeal mask airway insertion will take place. As per standard of care, an attending physician who is expert in pediatric airway management will supervise the procedure and intervene before the patient experiences excessive oxygen desaturation.

Apneic oxygenation will not be used as a long-term oxygenation strategy. No patient will be allowed to become hypoxic for research reasons.

All intubation procedures in both study groups will proceed as per usual practice. The goal of all intubation procedures has always been and remains the maintenance of adequate oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients presenting for surgery at University of New Mexico Children's Hospital
* Age range: adjusted gestational age 40 weeks, to 8 years

Exclusion Criteria:

* Patients whose airways would be maintained with mask ventilation only
* American Society of Anesthesiologists classes 4-6

Ages: 1 Day to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2015-05; Primary Completion 2018-03 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Codruta Soneru, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Children's Hospital, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- With-Cannula Group: Airway management (intubation) undertaken immediately after anesthetic induction, with simultaneous supplemental oxygen via nasal cannula.
  Supplemental oxygen via nasal cannula
Period: Overall Study
Arm/Group | Baseline Group | With-Cannula Group
Started | 200 | 160
Completed | 196 | 160
Not Completed | 4 | 0
Not completed — Protocol Violation | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline Group | With-Cannula Group | Total
Number analyzed (Participants) | 196 | 160 | 356
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 196 | 160 | 356
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3 [1.5 to 5] | 2 [1.2 to 4] | 3 [1.4 to 5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 67 | 154
  Male | 109 | 93 | 202
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 196 | 160 | 356
Weight [Median (Inter-Quartile Range); unit: kilograms] | 13.9 [10.4 to 19] | 13.4 [9.3 to 17.5] | 13.6 [10 to 18.4]
Height [Median (Inter-Quartile Range); unit: centimeters] | 95.3 [78.5 to 113] | 89.3 [73 to 107.8] | 92.5 [76 to 110.9]
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 16.6 [14.7 to 18.0] | 16.3 [14.9 to 18.1] | 16.4 [14.8 to 18.1]

OUTCOME MEASURES:

1. Primary Outcome: Time to First Event: Pulse Oximetry at 95%, or Successful Intubation
Description: Prior to anesthesia induction, patients are ventilated to achieve pulse oximetry (SpO2) values near 100%. This outcome represents the elapsed time before successful intubation or pulse oximetry declining to 95%, whichever came first.
Time Frame: From anesthetic induction to whichever comes first: pulse oximetry falling to 95%, or successful intubation; an expected average of less than 10 minutes
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Baseline Group | With-Cannula Group
Number analyzed (Participants) | 196 | 160
seconds | 106 [75 to 147] | 169 [128 to 225]

2. Secondary Outcome: Number of Patients Whose Pulse Oximetry Falls Below 95% During Airway Placement
Time Frame: From anesthetic induction to intubation; an expected average of 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Group | With-Cannula Group
Number analyzed (Participants) | 196 | 160
Participants | 85 | 14

3. Secondary Outcome: Number of Patients Requiring Intervention by Attending or Temporary Mask Ventilation During Airway Placement
Time Frame: From anesthetic induction to intubation; an expected average of 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Group | With-Cannula Group
Number analyzed (Participants) | 196 | 160
Participants | 52 | 22

4. Secondary Outcome: Number of Patients Whose Pulse Oximetry Falls Below 90% During Airway Placement
Time Frame: From anesthetic induction to intubation; an expected average of 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Group | With-Cannula Group
Number analyzed (Participants) | 196 | 160
Participants | 61 | 7

5. Secondary Outcome: Patients' Lowest Pulse Oximetry Value Observed During Airway Placement
Time Frame: From anesthetic induction to intubation; an expected average of 10 minutes
Measure: Median (Inter-Quartile Range); unit: percentage of oxygenated hemoglobin
Arm/Group | Baseline Group | With-Cannula Group
Number analyzed (Participants) | 196 | 160
percentage of oxygenated hemoglobin | 97 [89 to 99] | 99 [98 to 100]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the perioperative period: one day
Arm/Group | Baseline Group | With-Cannula Group
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/160
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/160
Other Adverse Events (participants affected / at risk) | 0/200 | 0/160

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT02437864/Prot_SAP_000.pdf